CLINICAL TRIAL: NCT07205432
Title: A Randomized, Double-blind, Placebo-controlled Phase I Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) Administration of XTL6001 Injection in Healthy and Obese Subjects
Brief Title: Phase I Study of XTL6001 Injection in Healthy and Obese Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Xitaili Biomedicine Technology co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XTL6001-I-C01
Record Dates: First submitted 2025-07-28; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-04

CONDITIONS: Weight Management in Adult Patients With Obesity or Overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XTL6001 (Experimental): Interventional: The SAD study involves single administration of XLT6001, while the MAD study involves administration of XLT6001 for no more than 4 weeks.
  Interventions: Drug: XTL6001
- Placebo (Placebo Comparator): Placebo: The SAD study involves single administration of Placebo, while the MAD study involves administration of Placebo for no more than 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XTL6001 — XTL6001 is a triple-target Glucagon-like peptide-1 receptor （GLP-1R） relevant agonist, intending to manage overweight/obesity and other metabolic diseases
  Arms: XTL6001
Drug: Placebo — This intervention contains no active ingredients
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled Phase I study to evaluate safety, PK and PD of single ascending dose (SAD) and multiple ascending dose (MAD) of XTL6001 injection in healthy and obese adult subjects.

SAD study: Includes 5 dose cohorts, with 40 subjects planned for enrollment. MAD study Includes 2 dose cohorts, with 30 subjects planned for enrollment.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Subjects in SAD part:

1. Age ≥ 18 and < 65 years at screening.
2. Body mass index (BMI) ≥ 18.5 kg/m² and < 28.0 kg/m² at screening.
3. Body weight ≥ 50.0 kg for males and ≥ 45.0 kg for females at screening.
4. Signed informed consent form prior to the trial, with full understanding of the study objectives, procedures, and potential adverse reactions.

Inclusion Criteria for Subjects in MAD part:

1. Age ≥ 18 and < 65 years at screening.
2. BMI ≥ 18.5 kg/m2且 < 40.0kg/m².
3. Body weight ≥ 50.0 kg for males and ≥ 45.0 kg for females at screening.
4. Stable body weight (fluctuation < 5%) for at least 3 months prior to screening.
5. Signed informed consent form prior to the trial, with full understanding of the study objectives, procedures, and potential adverse reactions.

Exclusion Criteria:

Exclusion Criteria for Subjects in SAD part:

1. History of type 1 or type 2 diabetes mellitus, or HbA1c > 6.5% or fasting plasma glucose > 7.0 mmol/L at screening.
2. Clinically significant gastric emptying disorders, chronic use of medications directly affecting gastrointestinal motility, severe chronic gastrointestinal diseases, or prior gastrointestinal surgery.
3. History of acute or chronic pancreatitis.
4. Symptomatic gallbladder disease.
5. Malignancy within 5 years prior to screening (except adequately treated non-melanoma skin cancer).
6. Personal/family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2A/2B (MEN 2A/2B).
7. Female subjects with positive pregnancy test or lactation.

Exclusion Criteria for Subjects in MAD part:

1. History of type 1 or type 2 diabetes mellitus, or HbA1c > 6.5% or fasting plasma glucose > 7.0 mmol/L at screening.
2. UnderlyingCushing's syndrome, hypothyroidism, PCOS,.
3. Clinically significant gastric emptying disorders, chronic use of medications directly affecting gastrointestinal motility, severe chronic gastrointestinal diseases, or gastrointestinal surgeries that may compromise safety or data interpretation.
4. History of acute or chronic pancreatitis.
5. Symptomatic gallbladder disease.
6. Malignancy within 5 years prior to screening (except adequately treated non-melanoma skin cancer).
7. Personal/family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2A/2B (MEN 2A/2B).
8. Female subjects with positive pregnancy test or lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of AEs (Adverse Events) and SAEs (Serious Adverse Events) | SAD: up to Day 8 MAD: up to Day 57

SECONDARY OUTCOMES:
The maximum plasma concentration (Cmax) of XTL6001 | Within 1 hour before each weekly dosing, and at 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168 hours after the first and last dose administration of the target dose level.
  Cmax - Maximum plasma concentration
Tmax of XTL6001 | Within 1 hour before each weekly dosing, and at 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168 hours after the first and last dose administration of the target dose level.
  The time to maximum concentration (Tmax) of XTL6001
Elimination half-life (T1/2) of XTL6001 | Within 1 hour before each weekly dosing, and at 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168 hours after the first and last dose administration of the target dose level.
  t1/2 - Elimination half-life
Area under the plasma concentration-time curve during one dosing interval (AUC) 0-tau of XTL6001 | Within 1 hour before each weekly dosing, and at 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168 hours after the first and last dose administration of the target dose level.
  AUC0-tau - Area under the plasma concentration-time curve during one dosing interval
AUC0-t of XTL6001 | Within 1 hour before each weekly dosing, and at 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168 hours after the first and last dose administration of the target dose level.
  AUC0-t - Area under the plasma concentration-time curve from time zero to the last measurable concentration
Body weight | MAD: up to Day57
  Body weight
Body mass index （BMI） | MAD: up to Day57
  Body mass index
Waist circumference | MAD: up to Day57
  waist circumference
Waist-to-hip ratio | MAD: up to Day57
  waist-to-hip ratio
Blood lipids | MAD: up to Day57
  Total cholesterol, triglycerides, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, apolipoprotein A1 and apolipoprotein B
Blood glucose | MAD: up to Day57
  Blood glucose
Insulin | MAD: up to Day57
  Insulin
Uric acid | MAD: up to Day57
  Uric acid
Anti-drug antibodies (ADA) | MAD: up to Day57
  Incidence of anti-drug antibodies (ADA)
ADA | MAD: up to D57
  Time to ADA positivity

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Shijitan Hospital, Capital Medical University, Beijing, Beijing Municipality, China